CLINICAL TRIAL: NCT02555280
Title: A 2 and 5 Year Evaluation of Clinical Outcomes in the Treatment of Degenerative Spinal Stenosis With Concomitant Low Back Pain by Decompression With Additional Stabilization Using the Coflex® Interlaminar Technology for FDA Actual Conditions for Use Study.
Brief Title: Coflex PS3 Actual Conditions for Use Study
Acronym: PAS003
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xtant Medical (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS3/P110008
Record Dates: First submitted 2015-09-02; First posted 2015-09-21 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Spinal Stenosis Lumbar
Keywords: moderate lumbar stenosis; neurogenic claudication; spinal stenosis; low back pain; decompression
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain | interventions — Decompression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- The coflex® Interlaminar Technology (Other): The coflex device was designed to address the clinical needs of spinal stenosis patients by providing stabilization of the affected level without fusion. The coflex is an interspinous process functional dynamic implant designed to impart a stabilizing effect at the treated level(s). The coflex device was approved by FDA in 2012.
  Interventions: Device: coflex® Interlaminar Technology
- Decompression (Active Comparator): Lumbar decompression back surgery is when a small portion of the bone over the nerve root and/or disc material from under the nerve root is removed to give the nerve root more space and provide a better healing environment.
  Interventions: Procedure: Decompression

INTERVENTIONS:
Device: coflex® Interlaminar Technology — Decompression plus coflex® Interlaminar Technology
  Other Names: coflex
  Arms: The coflex® Interlaminar Technology
Procedure: Decompression — Decompression alone
  Arms: Decompression

SUMMARY:
A 2 and 5 year evaluation of clinical outcomes in the treatment of degenerative spinal stenosis with concomitant low back pain by decompression with additional stabilization using the coflex® Interlaminar Technology for FDA Actual Conditions of Use Study.

DETAILED DESCRIPTION:
A prospective, multi center, concurrently enrolled, propensity score controlled through Month 60. The purpose is to fully characterize safety and efficacy then the coflex device is used in the intended subject population under actual conditions of use.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographic confirmation of at least moderate lumbar stenosis at one or two contiguous levels from L1-L5 that require surgical decompression.
2. Visual Analog Scale back pain score of at least 50 mm on a 100 mm scale.
3. Neurogenic claudication as defined by leg/buttocks or groin pain that can be relieved by flexion such as sitting in a chair.
4. Subject has undergone at least one lumbar injection at any prior time point, AND/OR at least 6 months of prior conservative care without adequate and sustained symptom relief.
5. Skeletally mature
6. Oswestry Low Back Pain Disability Questionnaire score of at least 20/50 (40%).
7. Psychosocially, mentally, and physically able to fully comply with this protocol, including adhering to scheduled visits, treatment plan, completing forms, and other study procedures.
8. Personally signed and dated informed consent document prior to any study-related procedures indicating that the patient has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

1. Prior fusion or decompressive laminectomy at index lumbar level.
2. Radiographically compromised vertebral bodies at any lumbar level(s) caused by current or past trauma or tumor (e.g., compression fracture).
3. Severe facet hypertrophy that requires extensive bone removal which would cause instability.
4. Isthmic spondylolisthesis or spondylolysis (pars fracture).
5. Degenerative lumbar scoliosis (Cobb angle of greater than 25°).
6. Osteoporsis or is at increased risk of osteoporosis.
7. Back or leg pain of unknown etiology.
8. Axial back pain only, with no leg, buttock, or groin pain.
9. Morbid obesity defined as a body mass index > 40.
10. Known allergy to titanium, titanium alloys, or MR contrast agents.
11. Active or chronic infection - systemic or local.
12. Cauda equina syndrome, defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder (bladder retention or incontinence) dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
coflex performance compared to IDE | 24and 60 Months
  Evaluation of coflex device performance in conjunction with surgical decompression in an actual conditions of use study.
coflex performance compared to decompression alone from ESCADA study. | 24 Months
  To compare clinical status of patients implanted with the coflex device in conjunction with surgical decompression relative to surgical decompression alone from ESCADA study.
Composite Clinical Success (CCS) | 24 Month
  * No secondary surgical interventions
  * No lumbar epidural injection, nerve block procedures at index level to treat spinal stenosis at any lumbar level
  * 15 point improvement in ODI in subjects with no interventions or injections
  * No new or increasing sensor or motor deficit
  * No major device related adverse events

SECONDARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | Baseline, 24 and 60 months
  Quality of life as determined by ODI. In terms of achieving at least a 15 point improvement.
Change in Visual Analog Scale (VAS) for low back pain | Baseline, 24 and 60 Months
  Low back pain reduction evaluated by use of VAS for back pain. In terms of achieving at least a 20 point improvement.
Change in Visual Analog Scale (VAS) for leg pain | Baseline, 24 and 60 Months
  Leg pain reduction evaluated by use of VAS for leg pain. In terms of achieving at least a 20 point improvement.
Neurological Status | Baseline, 6 weeks, 12, 24, 36, 48, 60 Months
  Assessment of maintenance of improvement after surgery.
Radiographic Assessments | 6 weeks, 12, 24, 60 Months
  * Significant migration or complete expulsion of implant
  * Spinous process fracture
  * Maintenance of foraminal height
  * adjacent level disease
Modified CCS | 24 Month
  CCS will be modified to include no use of a narcotic (opioids or opiates).
Medication Usage | 24 Month
  No use of narcotic (opioids and/or opiates)

OTHER OUTCOMES:
Safety Evaluation | Procedure, 6 week, 12, 24, 36, 48, 60 Months
  Safety will be evaluated by assessing the incidence of device and/or procedure related adverse events, revision, additional stabilizations

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Desert Institute for Spine Care (DISC), Phoenix, Arizona
  - Hoag Orthopedics, Irvine, California
  - Sutter Health, Sacramento, California
  - Central Cost Neurological Surgery, San Luis Obispo, California
  - Cervical Disc Center of Los Angeles, Santa Monica, California
  - UC Health Spine Center, Aurora, Colorado
  - Mercy Regional Medical Center, Durango, Colorado
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - 01L_Northshore University Health System, Evanston, Illinois
  - 24_Unity Surgical Center, LLC, Lafayette, Indiana
  - Orthopaedic Specialist of Northwest Indiana, Munster, Indiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - St. Joseph's Medical Center, Wayne, New Jersey
  - Northwell Health Physician Partners Orthopaedic Institute at Great Neck, Great Neck, New York
  - Consulting Orthopaedic Associates, Toledo, Ohio
  - Southern Oregon Orthpaedics, Medford, Oregon
  - Summit Spine, Portland, Oregon
  - 03L_Thomas Jefferson University, Philadelphia, Pennsylvania
  - Austin Neurosurgeons, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02555280/Prot_SAP_000.pdf